CLINICAL TRIAL: NCT01735708
Title: Treating Chronic Pain and Depression in HIV+ Patients in Primary Care Settings
Acronym: HIVPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Brown University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Lisa Uebelacker, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NR13438; R21NR013438 (NIH)
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Pain Interference; Depression; Antiretroviral Adherence
Keywords: pain; depression; HIV; adherence
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Education (Placebo Comparator): Participants in the Health Education arm will receive 7 individual sessions, each of which will focus on a different health education topic.
  Interventions: Other: Health Education
- HIVPASS Intervention (Active Comparator): Participants in the HIVPASS intervention arm will receive 7 individual sessions with the study interventionist, the first of which is a collaborative meeting with the PCP. Sessions will focus on pain interference and depression management.
  Interventions: Behavioral: HIVPASS

INTERVENTIONS:
Behavioral: HIVPASS
  Arms: HIVPASS Intervention
Other: Health Education
  Arms: Health Education

SUMMARY:
The purpose of this study is to determine whether participation in the study intervention, which involves collaboration between the study interventionist and the participant's primary care physician, will reduce symptoms of pain and depression in HIV+ patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain (pain duration for at least six months with a mean score of 5 or higher on the BPI Pain Interference Scale)
* Pain severity of 40 or higher on a Visual Analog Scale (0-100) indicating "worst pain in the last week"
* At least one trial of PCP-recommended medication (i.e. acetominophen, NSAIDS, skeletal muscle relaxants) judged through interviews with patients and PCPs
* QIDS score of ≥ 9 (depression severity)
* Stable dose of an antidepressant, if using, for the previous 2 months
* Age 18 or older
* HIV+

Exclusion Criteria:

* Lifetime DSM-IV diagnosis of bipolar disorder, schizophrenia, or other chronic psychotic condition
* Current DSM-IV diagnosis of substance dependence for alcohol, sedative/ hypnotic drugs, stimulants, or cocaine
* Suicidal ideation or behavior requiring immediate attention
* In psychotherapy or in a multidisciplinary pain management program
* Expected surgery in the next 6 months
* Pain thought to be due to cancer, infection, or inflammatory arthritis
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Uebelacker LA, Weisberg RB, Herman DS, Bailey GL, Pinkston-Camp MM, Garnaat SL, Stein MD. Pilot Randomized Trial of Collaborative Behavioral Treatment for Chronic Pain and Depression in Persons Living with HIV/AIDS. AIDS Behav. 2016 Aug;20(8):1675-81. doi: 10.1007/s10461-016-1397-7. PMID 27115400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Education | HIVPASS Intervention
Started | 95 | 92
Month 3 Assessment | 79 | 79
Completed | 84 | 79
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Education | HIVPASS Intervention | Total
Number analyzed (Participants) | 95 | 92 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.4) | 51.7 (8.8) | 51.4 (10.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 37 | 43 | 80
  Gender: Male | 56 | 49 | 105
  Gender: Non-binary | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 83 | 79 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 34 | 27 | 61
  White | 37 | 35 | 72
  More than one race | 16 | 12 | 28
  Unknown or Not Reported | 5 | 11 | 16
Brief Pain Inventory - Interference Scale [Mean (Standard Deviation); unit: units on a scale] — Title: Brief Pain Inventory Interference Scale. Abbreviation: BPI-I. Measures: self-report of interference due to pain. Scale range: 0-10. Higher scores represent a worse outcome.
  units on a scale | 6.44 (2.15) | 6.16 (1.98) | 6.30 (1.56)
Worst pain severity, past week [Mean (Standard Deviation); unit: units on a scale] — Title: worst pain severity, past week. Measures: self-report of worst pain in the past week. Scale range: 0-10. Higher scores represent a worse outcome.
  units on a scale | 8.27 (1.52) | 8.14 (1.61) | 8.21 (2.07)
Average pain severity, past week [Mean (Standard Deviation); unit: units on a scale] — Title: average pain severity, past week. Measures: self-report of average pain level in the past week. Scale range: 0-10. Higher scores represent a worse outcome.
  units on a scale | 6.37 (1.88) | 6.48 (1.87) | 6.43 (1.87)
Quick Inventory of Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Quick Inventory of Depressive Symptoms. Abbreviation: QIDS. Measures: clinician-based assessment of depression symptom severity. Scale range: 0-27. Higher scores represent a worse outcome.
  units on a scale | 14.4 (2.93) | 14.0 (3.04) | 14.2 (2.99)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — Title: Patient-Reported Outcome Measurement Information System (PROMIS) Anxiety Scale.
  Abbreviation: PROMIS Anxiety. Measures: self-report of anxiety symptom severity. Scale range: 8-40. Higher scores represent a worse outcome.
  units on a scale | 24.5 (6.44) | 24.5 (6.63) | 24.5 (6.39)
Antiretroviral therapy (ART) adherence [Mean (Standard Deviation); unit: % Adherence] — Antiretroviral Therapy (ART) Adherence. Measures: self-report of percent adherence to ART within the past month. Range: 0-100%. Higher scores represent better adherence.
  % Adherence | 91.5 (18.4) | 95.1 (0.5) | 93.3 (15.1)
Detectable viral load [Count of Participants; unit: Participants] | 20 | 13 | 33
SF-36 Physical Health component [Mean (Standard Deviation); unit: units on a scale] — 36-item Short Form Survey -- Physical Health Component. Abbreviation: SF-36 Physical Health Component. Measures: quality of life related to physical health, via self-report. Range in this sample: -3.41 - 1.36. Higher scores represent better functioning.
  units on a scale | -1.67 (0.94) | -1.42 (1.07) | -1.55 (1.01)
SF-36 Mental Health component [Mean (Standard Deviation); unit: units on a scale] — 36-item Short Form Survey-- Mental Health Component. Abbreviation: SF-36 Mental Health Component. Measures: quality of life related to mental health, via self-report. Range in this sample: -4.48 - 1.36. Higher scores represent better functioning.
  units on a scale | -1.83 (1.09) | -1.77 (1.21) | -1.80 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory Interference Scale at 3 Months
Description: Title: Brief Pain Inventory Interference Scale. Abbreviation: BPI-I. Measures: self-report of interference due to pain. Scale range: 0-10. Higher scores represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education | HIVPASS Intervention
Number analyzed (Participants) | 79 | 79
score on a scale | 5.03 (2.98) | 4.23 (2.84)
Statistical Analysis 1: Comparison: Health Education vs HIVPASS Intervention; Test type: Superiority — ITT analysis using multiple imputation by chained equation with 50 fully populated data sets; p = 0.008, Mixed Models Analysis — A priori threshold for significance was two-tailed p = .05; Standard errors were based on robust Huber-White variance estimator; Mean Difference (Net) = -1.31, 95% CI 2-sided [-2.28 to -0.34], Standard Error of Mean 0.493 — standard error of difference in means

2. Secondary Outcome: Brief Pain Inventory Interference Scale at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education | HIVPASS Intervention
Number analyzed (Participants) | 84 | 79
score on a scale | 4.74 (3.12) | 4.95 (3.01)
Statistical Analysis 1: Comparison: Health Education vs HIVPASS Intervention; Test type: Superiority — Intent to treat analysis using multiple imputation by chained equations with 50 fully populated data sets; p = 0.251, Mixed Models Analysis — A priori threshold for significance was two-tailed p = .05; Standard errors were based on robust Huber-White variance estimator; Mean Difference (Net) = -0.57, 95% CI 2-sided [-1.53 to 0.40], Standard Error of Mean 0.495

3. Secondary Outcome: Quick Inventory of Depression Symptoms at 3 Months
Description: Quick Inventory of Depressive Symptoms. Abbreviation: QIDS. Measures: clinician-based assessment of depression symptom severity. Scale range: 0-27. Higher scores represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Health Education: Participants in the Health Education arm will receive 7 individual sessions, each of which will focus on a different health education topic.
  Health Education
- HIVPASS Intervention: Participants in the HIVPASS intervention arm will receive 7 individual sessions with the study interventionist, the first of which is a collaborative meeting with the PCP. Sessions will focus on pain interference and depression management.
  HIVPASS
Arm/Group | Health Education | HIVPASS Intervention
Number analyzed (Participants) | 79 | 79
score on a scale | 10.35 (4.81) | 10.25 (4.81)
Statistical Analysis 1: Comparison: Health Education vs HIVPASS Intervention; Test type: Superiority — Intent to treat analysis using multiple imputation by chained equations with 50 fully populated data sets; p = 0.844, Mixed Models Analysis — A priori threshold for significance was two-tailed p = .05; Standard errors were based on robust Huber-White variance estimator; Mean Difference (Net) = 0.15, 95% CI 2-sided [-1.32 to 1.61], Standard Error of Mean 0.750 — Standard error of difference in means

4. Secondary Outcome: Quick Inventory of Depression Symptoms at 12 Months
Description: as for outcome 3
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education | HIVPASS Intervention
Number analyzed (Participants) | 84 | 79
score on a scale | 10.18 (5.05) | 9.80 (5.60)
Statistical Analysis 1: Comparison: Health Education vs HIVPASS Intervention; Test type: Superiority — Intent to treat analysis using multiple imputation by chained equations with 50 fully populated data sets; p = 0.545, Mixed Models Analysis — A priori threshold for significance was two-tailed p = .05; Standard errors were based on robust Huber-White variance estimator; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-2.18 to 1.15], Standard Error of Mean 0.836 — Standard error of difference in means

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Health Education | HIVPASS Intervention
All-Cause Mortality (participants affected / at risk) | 2/95 | 2/92
Serious Adverse Events (participants affected / at risk) | 39/95 | 21/92
Other Adverse Events (participants affected / at risk) | 40/95 | 35/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Health Education (N=95) | HIVPASS Intervention (N=92)
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bacteremia (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chest pain (Cardiac disorders) | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Cranial nerve palsy (Eye disorders) | 0 | 1
Deep vein thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Detox (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Edema in limbs (General disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
GI bleed (Gastrointestinal disorders) | 1 | 1
Heart failure (Cardiac disorders) | 1 | 0
Hospitalization/reason unknown (General disorders) | 4 | 2
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Kidney infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 3
Meningitis (Infections and infestations) | 0 | 1
Nausea/vomiting/GI pain (Gastrointestinal disorders) | 2 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Otitis media externa (Infections and infestations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 2
Renal calculi (Renal and urinary disorders) | 0 | 1
Renal insufficiency (Renal and urinary disorders) | 1 | 1
Seizure (Nervous system disorders) | 4 | 0
Sepsis (Infections and infestations) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Suicide ideation (Psychiatric disorders) | 2 | 0
Surgical or medical procedure (Surgical and medical procedures) | 5 | 2
Syncope (Nervous system disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Health Education (N=95) | HIVPASS Intervention (N=92)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7
Fall (Injury, poisoning and procedural complications) | 10 | 6
Nausea, vomiting, and/or GI pain (Gastrointestinal disorders) | 9 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4
Surgical or medical procedure (Surgical and medical procedures) | 7 | 3
Upper respiratory infection (Infections and infestations) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No